CLINICAL TRIAL: NCT01162824
Title: Correlation Between Abnormal Coronary Vasoreactivity Testing, Expansion of CD4+CD28null T Cells and Biomarkers for Inflammation and Endothelial Dysfunction in Patients With Angina Despite Angiographically Normal Coronary Arteries.
Brief Title: Blood Markers for Inflammation and Coronary Artery Vasoreactivity Testing in Patients With Chest Pain and Normal Coronary Arteries
Acronym: ACOVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St George's Healthcare NHS Trust (Other)
Responsible Party: Professor JC Kaski, Department of Cardiology, St George's Healthcare NHS Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ACOVA-8
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Endothelial Dysfunction; Atherosclerosis; Inflammation; Myocardial Ischemia
Keywords: Endothelial Dysfunction; Microvascular dysfunction; Coronary artery spasm; Inflammation; CD4+CD28null T cells; Myocardial ischemia; Early atherosclerosis
MeSH Terms: conditions — Atherosclerosis; Inflammation; Myocardial Ischemia; Coronary Vasospasm | interventions — Acetylcholine; lactitol; Adenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No endothelial dysfunction (Other)
  Interventions: Drug: Acetylcholine; Drug: Adenosine
- Endothelial Dysfunction (Other): Definition of abnormal epicardial and microvascular vasoreactivity Abnormal epicardial vasoreactivity is defined as a reduction of the baseline coronary diameter ≥75% after glyceryltrinitrate i.c. together with a reproduction of the angina symptoms reported by the patient and/or ischemic ECG-changes. Abnormal microvascular vasoreactivity is defined as the reproduction of the angina symptoms together with ischaemic ECG-changes, but without changes in epicardial vasomotion.
  Interventions: Drug: Acetylcholine; Drug: Adenosine

INTERVENTIONS:
Drug: Acetylcholine — Incremental doses of 2, 20 and 100 µg of ACH will be injected into the left coronary artery (LCA) via the diagnostic catheter for 3 minutes each. After that 80 µg of ACH will be injected into the right coronary artery. Coronary angiography will be performed after each 3 minute dose period. After the test or when intolerable chest pain due to coronary spasm occurs, 0.2 mg of glyceryltrinitrate will be injected into each vessel. During the test, heart rate, blood pressure and ECG will be monitored continuously.
  Other Names: Acetylcholine will be used from Miochol-E (Novartis)
Drug: Adenosine — Coronary blood flow velocity measurements will be performed in the mid segment of the left anterior descending artery with a 0.014-in intracoronary Doppler guidewire connected to the corresponding interface. Measurements will be obtained after the administration of nitroglycerin, at baseline and during maximal hyperaemia. Sustained intravenous administration of adenosine - an arteriolar vasodilator- will be used to induce maximal hyperaemia (140-180µg/kg/min).

SUMMARY:
The investigators are hoping to discover the cause of chest pain in patients with a normal coronary arteriogram. For patients with chest pain coronary angiography is the standard method by which the blood vessels of the heart can be visualized and any narrowing can be assessed. In some cases the investigators find totally normal coronary blood vessels or only minor disease. Such a finding is associated with an excellent long term prognosis. However, as a large proportion of patients with normal coronary arteries or mild coronary narrowings often continue to experience recurrent chest pains the investigators are interested in understanding the mechanisms responsible for this. The investigators hypothesise that in many cases, coronary artery spasms are responsible for the recurrent chest pains. These spasms usually respond to treatment with drugs known as vasodilators. The acetylcholine test (ACH-test) has been recommended by the European Society of Cardiology and the American College of Cardiology as a diagnostic test. This test can reveal whether the coronary blood vessels have a tendency to go into spasm. The investigators plan in this study to carry out the test in patients who have chest pains suggestive of coronary narrowings but are found to have normal or only mildly narrowed coronary arteries on angiography. A positive test -indicating a tendency for spasm- may help guiding therapy with vasodilators, which are often very effective to prevent coronary spasms. The investigators would also like to take blood samples during the test (before and after) from every patient to measure blood markers and see if there is a relation between these markers and the result of the ACH-test.

DETAILED DESCRIPTION:
This study comprises two parts:

1. Blood sample
2. ACH-test (including coronary flow measurements)

Blood will be taken, frozen and stored for up to 5 years. The following markers will be studied: C-reactive protein, E-selectin, neopterin, troponin and CD40 ligand. These are essential biochemical markers or so called pro-inflammatory substances that normally circulate in the blood but their levels can increase under certain conditions such as stress or inflammation. In addition, expansion of CD4+CD28null T-cells will be measured via flow cytometry.

Coronary angiography will be performed according to routine clinical guidelines. If the investigators find severe disease standard treatment procedures will take place and the investigators will only ask for a blood sample. If the investigators find normal coronary arteries on coronary angiography the investigators will conduct the ACH-test as part of the study. After injecting ACH into the coronary arteries narrowing can occur and provoke the same or similar symptoms as at home (i.e. chest pain). If you experience severe pain the investigators will inject a drug called nitroglycerine to relieve the pain. Then the investigators will measure the capacity of the blood vessels to dilate with a special catheter. The whole procedure including coronary angiography and ACH-test will last for about one hour. There is only very little radiation needed for the ACH-test which is unlikely to cause any health problems (~2.4mSv). In some very rare cases chest pain can be prolonged and heart rhythm disorders can occur. In worst case prolonged narrowing can lead to a heart attack (myocardial infarction, < 1%).

The result of the ACH-test can lead to 3 different results.

1. Epicardial coronary spasm. This means that the narrowing of the blood vessel occurs in a place where it can be seen on the screen during angiography.
2. Microvascular dysfunction This means that the narrowing of the blood vessel cannot be seen on the screen but on the ECG. It only affects the very small blood vessels of the heart.
3. Normal ACH-test This means that the test is normal and the patient has no chest pain during the test and also no narrowing.

Depending on the result the investigators will suggest to start with a medication according to current guidelines and inform the patient's GP about the results and further suggestions for treatment. To maintain confidentiality all participants are entered onto our secure database using only their initials and a study number.

ELIGIBILITY:
Inclusion Criteria:

* Adults of either gender > 35 years of age with a stable pattern of angina pectoris suggestive of coronary artery disease, with positive responses to exercise stress testing AND/OR patients with chest pain and ischaemic ST-segment changes during pain (previous obstructive coronary artery disease with or without stent-implantation will be allowed).
* Subjects will be invited to participate only if investigations have been undertaken to rule out non-cardiac causes for chest pain (i.e. oesophageal and musculoskeletal) previously.
* Serum creatinine < 123.7µmol/L.
* Left ventricular ejection fraction > 50%.

Exclusion Criteria:

* Chronic obstructive pulmonary disease.
* Cardiomyopathy.
* Severe valvular heart disease.
* Myocardial infarction within the last 3 months.
* Pregnant or lactating women.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Endothelial Dysfunction | Day 1 (day of study entry)
  As this is not a follow-up study, the intracoronary vasoreactivity tests will be conducted at the day of study entry to assess which patient suffers from endothelial dysfunction. According to this result the patients will be divided into two groups (endothelial dysfunction and NO endothelial dysfunction).
  Definition of endothelial dysfunction:
  Vasoconstriction of >75% together with ischemic ECG changes and/or reproduction of angina OR ischemic ECG changes with reproduction of angina without vasoconstriction

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Kaski, MD, Principal Investigator — Department of Cardiology, St George's Healthcare NHS Trust
Locations (1):
- Department of Cardiology, St George's Healthcare NHS Trust, London, England, United Kingdom